CLINICAL TRIAL: NCT01979705
Title: A Prospective Study to Detect Novel Pathogens and Characterize Emerging Infections
Brief Title: Detect Novel Pathogens and Characterize Emerging Infections
Acronym: NP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NP 07/2013
Record Dates: First submitted 2013-10-30; First posted 2013-11-08 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Prospective Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood
  2. Throat Swab
  3. Nasal Swab
  4. ETT Swab (if patient is intubated)
  5. Urine
  6. Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infectious disease is the single biggest cause of death worldwide. New infectious agents,such as the Severe Acute Respiratory Syndrome coronavirus and new strains of influenza continually emerge and require new investigations to understand pathogen biology and pathogenesis in the host. Witness the Influenza A pandemic. Concerns about new viruses and their impact on health and the economy are also increasing. Current alerts sent out by the Ministry of Health (about the novel coronavirus and the Avian influenza A virus) are but cases in point. These likely reflect advances in science, which have allowed novel pathogens to be identified.

Because of its geography, Singapore is vulnerable to new pathogens through importation or the global travel of its citizens. Hence we must be ever ready to meet unexpected challenges anytime.

On the administrative front, Singapore General Hospital has a Disease Outbreak Task-force which has in place many plans that can be activated should there be a large-scale epidemic.

What is missing thus far is a program that will enable us to perform scientific studies in the setting of an epidemic. Hence in this study, we will, in collaboration with the Program in Emerging Infectious Diseases (EID) in Duke-National University of Singapore Postgraduate Medical School, attempt to (i) detect novel, previously undescribed pathogens; (ii) characterize viruses (not necessarily novel but emerging and re-emerging) that are raising concern or causing clusters or epidemics in the hospital and/or country; (iii) characterize immune responses to such viruses in healthcare workers as well as patients (those affected by these viruses and those exposed to the affected). The techniques that will be used will be those not routinely available in a hospital's service labs.

Some patients will remain undiagnosable with the best available technology. Since new laboratory tools that can detect previously undiagnosed pathogens may become available in the future, the study also aims to archive specimens from patients whose illnesses remain undiagnosed.

DETAILED DESCRIPTION:
This study has the following aims:

1. To detect novel, previously undescribed pathogens.
2. To characterize viruses (not necessarily novel but emerging and re-emerging) that are raising concern or causing clusters or epidemics in the hospital and/or country;
3. To characterize immune responses to such viruses in patients.
4. To archive specimens with no identifiable infectious etiological agents for future testing.

A recent global analysis documented that emerging infectious disease events have increased significantly over time. Singapore has not been spared with the list of pathogens since the late 1990s, including Nipahn virus, SARS coronavirus, dengue, chikungunya, and 2009 H1N1. As is widely known, the novel coronavirus may potentially impact Singapore as Haj pilgrims from Singapore travel to Saudi Arabia and are potentially exposed to this virus.

Novel pathogens continue to be discovered. An example of this is the Severe Fever with Thrombocytopenia Syndrome bunyavirus in Henan, China. Appropriately a commentary accompanying the report identified China as a country with the largest potential for emerging or re-emerging infectious disease, due to the close proximity of animals and human populations. Similarly, Southeast Asia was identified as a potential hotspot, citing the avian influenza pandemic and Nipahn virus outbreak. As such, it is obvious that there is a need to better define undiagnosed infective syndromes in Singapore, and subsequently characterize emerging pathogens.

In Singapore, there is currently a lack of research focus on discovery of novel pathogens. Our current protocol is an attempt to fill this gap. This proposal brings together experts in clinical infectious diseases in SGH, world renowned scientists in laboratory diagnostics of infectious diseases and public health epidemiology experts in Duke-NUS Postgraduate Medical School. We hope by employing state of the art technologies, we will be at the frontier of new pathogen discovery.

ELIGIBILITY:
Inclusion Criteria:

Any person admitted to Singapore General Hospital or seen as an outpatient in the Specialist Outpatient Clinic who has:

1. clinical history and/or clinical syndromes compatible with a suspected novel/re-emerging infective etiological agent

Exclusion Criteria:

1. Any person unable to give informed consent and for whom no legally acceptable representative is available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a prospective study with inclusion criteria as specified below:
  Inclusion criteria:
  Any person admitted to Singapore General Hospital or seen as an outpatient in the Specialist Outpatient Clinic who has:
  1. clinical history and/or clinical syndromes compatible with a suspected novel/re-emerging infective etiological agent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-08 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Detecting of Novel Pathogens | Day 1 - Day 28 of recruitment
  1. Clinical data collection through case records, and interview of patients or next-of-kin or friend in the event information is unavailable or incompletely documented in the case records.
  2. Sample collection will be performed according to the following frequency:
     1. First day of enrolment: blood draw (by weight) not more than 20ml, nasal (and/or nasopharyngeal ) and/or throat swab, stool and urine sample.
     2. On days 2, 3, 5, 7, 10, 14 and 28: blood (by weight) not more than 10 ml, nasal (and/or nasopharyngeal l) and/or throat swab, stool and urine sample. On D28, blood (by weight) not more than 20ml, will be drawn as most immune response changes manifest by then.
  If available, urine and stool sample will be collected. If the subject is intubated, endotracheal aspirate will replace nasal and throat swab. Sample collection for research will be done at the same time as samples for clinical testing as far as possible, to minimize patient discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Tan Ban Hock, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided